CLINICAL TRIAL: NCT07320898
Title: The Effect of Injectable Platelet-Rich Fibrin Application on Alkaline Phosphatase and MMP-9 Levels in Periapical Exudate and Gingival Crevicular Fluid of Teeth With Apical Periodontitis
Brief Title: Effect of I-PRF Application on ALP and MMP-9 Levels in Teeth With Apical Periodontitis
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Ali Turkyilmaz, Associate Professor, Kırıkkale University
Other Study IDs: 2024/17 - 2024.12.22
Record Dates: First submitted 2025-11-27; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Apical Periodontitis; i-PRF; Biomarkers; MMP-9; Alkaline Phosphatase
Keywords: apical periodontitis; Injectable platelet-rich fibrin; Alkaline phosphatase; Matrix metalloproteinase-9
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: 30 participants. Procedure: Root canal treatment without i-PRF application. Collection of GCF and PAE samples.
- I-PRF Group: 30 participants. Procedure: i-PRF application and root canal treatment. Collection of GCF and PAE samples.

SUMMARY:
The aim of this study was to evaluate the effect of injectable platelet rich fibrin (i-PRF) injection, in addition to routine root canal treatment, on alkaline phosphatase (ALP) and matrix metalloproteinase-9 (MMP-9) levels in teeth with chronic apical periodontitis. A total of 60 patients were included and randomly divided into two groups: the control group and the experimental group (i-PRF). Gingival crevicular fluid (GCF) samples and periapical exudate (PAE) samples were collected from the teeth at the first appointment, after completion of chemomechanical preparation. In both groups, calcium hydroxide was placed in the root canals, and the teeth were temporarily sealed with composite resin. While no additional procedure was performed in the control group, patients in the experimental group received submucosal i-PRF injection. The second samples were obtained after 4 weeks, and in the same session, the root canal treatment was completed, followed by permanent restoration. ALP and MMP-9 levels in the collected samples were analyzed using the ELISA test.

DETAILED DESCRIPTION:
The study was conducted with 60 volunteer patients aged 18-64, classified as ASA I, who presented to the Department of Endodontics at the Faculty of Dentistry, Kırıkkale University. They had chronic apical periodontitis in the upper or lower jaw and a periapical lesion diameter of less than 1 cm on either incisor or premolar. Before starting root canal treatment, GCF samples were collected from the included teeth. Plaque on the tooth surface from which GCF samples were to be collected was removed with cotton pellets, and then isolated with a cotton roll. The teeth were dried with compressed air. Paper strips were inserted into the pocket from the mesiobuccal and distobuccal surfaces of the tooth. They were advanced until pressure was felt at the pocket base. GCF was collected by holding the paper strips in the sulcus for 30 seconds. The GCF volume of the paper strips was measured using a Periotron 8000 device, and the researcher recorded the volumes. Paper strips contaminated with blood or saliva were excluded from the study. The paper strips included in the study were placed in Eppendorf tubes and stored at -20°C, then at -80°C, until the ELISA experiments were performed.

Sterile paper points were used to collect periapical exudate samples from teeth after the shaping and irrigation protocols were completed. The root canals were dried to the working length using a #40 paper point. The #20 paper points, adjusted to a length 2 mm longer than the working length, were moved 2 mm from the apical stop and held for 1 minute. The process was repeated three times. A 4-mm cut was made at the ends of the periapical exudate-impregnated paper points with sterile surgical scissors, and the resulting segments were transferred to the Eppendorf tubes. After collecting the periapical sample, calcium hydroxide paste was placed in the canal. The tooth was temporarily sealed with composite resin to prevent contamination between sessions.

The procedures described above were performed identically in both groups. In the i-PRF group, five cc of blood was collected from the patients' antecubital vein into a glass-coated plastic tube without anticoagulant. I-PRF was centrifuged at 700 rpm for 3 minutes. After centrifugation, the i-PRF obtained at the top of the tube was collected using a syringe. The canal length measured during treatment was used to apply i-PRF at the point closest to the tooth apex. To ensure standardization across all patients, 0.5 cc of i-PRF was injected submucosally at the designated site. In the second session, following isolation and disinfection as described in the first session, GCF samples were collected, and after the final irrigation procedure, PAE samples were collected. The root canals were obturated by the lateral condensation method using gutta-percha cones and root canal sealer. Permanent restorations were made with composite resin. The samples were analyzed with ELISA. Data analysis was performed using SPSS 27.0, and a 95% confidence level was achieved. Frequency and percentage (n (%)) are given for categorical (qualitative) variables, while mean, standard deviation, minimum, maximum, and median values are given for numerical (quantitative) variables. The dependent-samples t-test and the Wilcoxon test were used for repeated measurements in the study. The independent-samples t-test and Mann-Whitney U test were used to compare groups. The Spearman correlation test was used for relationships between measurements.

ELIGIBILITY:
Inclusion Criteria:

* Sixty patients who applied to Kırıkkale University Faculty of Dentistry and were diagnosed with chronic apical periodontitis and were included in the PAI 3-4 groups according to the Periapical Index Scoring System (PAI) among the patients who were prescribed root canal treatment were included in the study.
* Patients aged 18-64
* Upper or lower incisors and premolars with primary apical periodontitis
* Patients with ASA I
* Patients who have provided written informed consent to participate in the study.

Exclusion Criteria:

* Patients with ASA II or higher,
* Patients who have used antibiotics and anti-inflammatory medications within the last month,
* Patients with a periodontal pocket greater than 3 mm in the affected tooth,
* Teeth with internal or external root resorption, or teeth with swelling and pain on palpation,
* Pregnant women or those suspected of pregnancy,
* Patients with generalized periodontitis,
* Patients with immunosuppressive systemic diseases such as diabetes and hepatitis will not be included in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients between the ages of 18-64 years old and diagnosed with apical periodontitis who applied to Kırıkkale University, Faculty of Dentistry, Department of Endodontics with the indication of root canal treatment will be included in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
ALP and MMP-9 Levels in Periapical Exudate (PAE) and Gingival Crevicular Fluid (GCF) | Baseline and 28. Days
  In teeth with apical periodontitis, periapical exudate (PAE) and gingival crevicular fluid (GCF) collected during the first and second sessions of root canal treatment will be analyzed to measure alkaline phosphatase (ALP) and matrix metalloproteinase-9 (MMP-9) levels. ALP levels will be expressed in U/L, while MMP-9 levels will be expressed in ng/dL, and each enzyme will be measured and reported separately. Enzyme levels will be compared between the group receiving injectable platelet-rich fibrin (i-PRF) and the group not receiving i-PRF.

SECONDARY OUTCOMES:
Comparison of ALP and MMP-9 Levels Between Sessions and Sample Types | Baseline and 28. Days
  The secondary outcome will evaluate the differences in ALP and MMP-9 levels between the first and second sessions, and between the PAE and GCF samples. ALP values will be evaluated in U/L, and MMP-9 values in ng/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze E NALBANT, Research Assistant, Principal Investigator — Kirikkale University Faculty of Dentistry; Ali Türkyılmaz, Associate Professor, Study Chair — Kirikkale University Faculty of Dentistry
Locations (1):
- Kırıkkale University, Faculty of Dentistry, Kırıkkale, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided